CLINICAL TRIAL: NCT03729128
Title: The Potential Therapeutic Effects of add-on Low Dose Dextromethorphan and Memantine in Patients With Amphetamine-type Stimulants Use Disorder
Brief Title: Add-on Low Dose Dextromethorphan and Memantine in Patients With Amphetamine-type Stimulants Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tzu-Yun Wang (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Tzu-Yun Wang, Principal Investigator, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-BR-106-094
Record Dates: First submitted 2018-07-15; First posted 2018-11-02 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Stimulants Use Disorder
Keywords: amphetamine-type stimulants use disorder; dextromethorphan; memantine; inflammation; neurodegeneration
MeSH Terms: conditions — Inflammation; Nerve Degeneration | interventions — Dextromethorphan; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dextromethorphan and memantine (DM+MM) (Experimental): The patients with Amphetamine-type stimulants use disorder will be recruited and received treatment of add-on dextromethorphan 30mg/day and memantine 5mg/day combination (DM+MM) for 12 weeks.
  Interventions: Drug: dextromethorphan and memantine (DM+MM)
- Placebos (Placebo Comparator): The patients with Amphetamine-type stimulants use disorder will be recruited and received treatment of add-on placebos for 12 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: dextromethorphan and memantine (DM+MM) — Patients of Amphetamine-type stimulants use disorder (ATSUD) will take dextromethorphan 30 mg/day and memantine 5 mg/day combination (DM+MM) daily for 12 weeks.
  Arms: dextromethorphan and memantine (DM+MM)
Drug: Placebos — Patients of Amphetamine-type stimulants use disorder (ATSUD) will take placebos daily for 12 weeks.
  Arms: Placebos

SUMMARY:
The current study will investigate whether add-on dextromethorphan (DM) and memantine (MM) is able to improve the treatment outcomes for ATSUD, and be associated with improvement in inflammatory markers, neurotrophic factors and neuropsychological tests.

DETAILED DESCRIPTION:
In current study, we will conduct a randomized double-blind placebo-controlled study. We will recruit 100-120 patients with ATSUD in three years and allocate them to add-on low dose dextromethorphan and memantine (DM 30mg/day+MM 5mg/day) or placebo group in a 1: 1 ratio (patients will also undergo usual psychosocial interventions). We will follow up the participants for 12 weeks and measure the treatment responses, urine drug tests, craving scales and side effects to evaluate the therapeutic effects of add-on DM+MM. Neuropsychological assessments and tests for inflammatory parameters and neurotrophic factors will also be measured during 12-weeks follow up. The study results will show that whether add-on DM+MM is able to improve the treatment outcomes for ATSUD, and be associated with improvement in inflammatory markers, neurotrophic factors and neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of these inclusion criteria to be eligible for enrollment into the study:

1. Signed informed consent by patient or legal representative.
2. Male or female patient aged ≧20 and ≦65 years.
3. A diagnosis of ATSUD according to DSM criteria made by a specialist in psychiatry.
4. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

1. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study.
2. Females who are pregnant or lactation.
3. Other major Axis-I DSM-IV diagnosis other than ATSUD, except for tobacco use disorder, ATS induced mood or psychotic disorders.
4. Current evidence of an uncontrolled and/or clinically significant medical condition, e.g., cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation.
5. History of allergy or intolerable side effects of DM or MM.
6. Suicidal attempts or risks during screen or study period.
7. Presence of active infectious or autoimmune disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Urinary amphetamine tests | 12 weeks
  The urinary amphetamine tests will be examined during the 12 weeks of treatment period in patients with ATSUD and the results will be compared between the experimental and placebo groups.
Craving severity | 12 weeks
  The Visual analog scale (VAS) will be measured during the 12 weeks of treatment period in patients with ATSUD. The results will be compared between the experimental and placebo groups. The level of conscious craving was rated from 0 (none) to 100 (very much). Higher scores indicate more severe craving.
Side effects checklists | 12 weeks
  The investigators will use the self-reported questionnaire, side effects checklists, to evaluate the side effects during the 12 weeks of treatment period in patients with ATSUD. The side effects assessment includes, A) Mental Status/6-item, B) Genito-Urinary/4-item, C) Cardiovascular/4-item, D) Head-Neck/10-item, E) Extremities/9-item, F) Skin/4-item, and G) Gastrointestinal Tract/2-item. The severity of side effects were divided into 4 degrees as follows: 0 = Not present; 1 = Mild or occasional; 2 = Moderate or occurs several times a day; and 3 = Severe or persistent. Scores in each subscale will be summated to get the final total scores. Higher scores indicate more severe side effects. The results of side effects checklists will be compared between the experimental and placebo group.

SECONDARY OUTCOMES:
Wisconsin Card Sorting Test (WCST) | 12 weeks
  The Wisconsin Card Sorting Test (WCST) will be measured in patients with ATSUD at the initial screen period and at the endpoint (after 12 weeks of treatment). We will compare the changes from screen period to the endpoint between experimental and placebo group. Performance on the WCST was scored in terms of the total number of errors (TNE, range form 0-128), perseverative errors (PE, range from 0-118), conceptual level responses (CLRs, range from 0-100%), number of categories completed (NCC, range form 0-12), and trials to complete the first category (TCC, range from 0-128). Higher scores indicate worse performance in TNE, PE, and TCC. Higher scores indicate better performance in CLRs and NCC.
Continuous performance tests (CPT) | 12 weeks
  The Continuous performance tests (CPT) will be measured in patients with ATSUD at the initial screen period and at the endpoint (after 12 weeks of treatment). We will compare the changes from screen period to the endpoint between experimental and placebo group. The CPT produces a standard set of performance measures that include the number of errors of omission and errors of commission. (1) Errors of omission occur when the participant fails to respond to the target stimulus. The omission errors t-scores are ranged from 20-80 (0-100%). Higher scores indicated worse performance. (2) Errors of commission occur when the participant responds to a non-target (X) stimulus. The commission errors t-scores are ranged from 20-80 (0-100%). Higher scores indicated worse performance.
Wechsler Memory Scale - third edition (WMS-III) | 12 weeks
  The Wechsler Memory Scale - third edition (WMS-III) will be measured in patients with ATSUD at the initial screen period and at the endpoint (after 12 weeks of treatment). We will compare the changes from screen period to the endpoint between experimental and placebo group. WMS-III composite scores were calculated for the eight standardized primary indices: Auditory Immediate (AIM, range from 50-156), Visual Immediate (VIM, range from 47-162 ), Immediate Memory (IM, range from 40-164 ), Auditory Delayed (ADM, range from 46-162), Visual Delayed (VDM, range from 43-156), Auditory Recognition Delayed (ARDM, range from 55-145), General Memory (GM, range from 40-168), and Working Memory (WM, range from 45-156 ). Higher scores indicate better performance.
Cytokines and neurotrophic factors | 12 weeks
  The plasma levels of cytokines and neurotrophic factors, tumor necrosis factor α (TNF-α[pg/mL]), transforming growth factor β1 (TGF-β1 [pg/mL]), interleukin 6( IL-6[pg/mL]), interleukin 8(IL-8[pg/mL]), interleukin 1β (IL-1β[pg/mL]), and brain-derived neurotrophic factor(BDNF[pg/mL]), will be measured in patients with ATSUD at the initial screen period, day 1(baseline), week 4, 8, and 12(endpoint). We will compare the changes from screen period to the endpoint between the experimental and placebo group.
C-reactive protein | 12 weeks
  The plasma levels of C-reactive protein (CRP[μg/mL]) will be measured in patients with ATSUD at the initial screen period, day 1(baseline), week 4, 8, and 12(endpoint). We will compare the changes from screen period to the endpoint between the experimental and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yun Wang, Principal Investigator — National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan